CLINICAL TRIAL: NCT04137627
Title: Effect of Melatonin in Combination With Neoadjuvant Chemotherapy to HIF-1⍺, CD44, CD133, and miR-210 Expression and Clinical Response in Locally Advanced Oral Squamous Cell Carcinoma (OSCC)
Brief Title: Melatonin Effect in Combination With Neoadjuvant Chemotherapy to Clinical Response in Locally Advanced Oral Squamous Cell Carcinoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Diani Kartini,SpB(K)Onk, Lecturer, Staff of Oncology Division of Department of Surgery, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: MLTOSCC
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Oral Squamous Cell Carcinoma; Neoadjuvant Chemotherapy
Keywords: Melatonin; Locally Advanced Oral Squamous Cell Carcinoma; Neoadjuvant Chemotherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Melatonin

STUDY DESIGN:
Intervention Model Description: one group receive standard treatment with melatonin, while the other group receive standard treatment with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Melatonin (Experimental): The group received standard treatment with the oral administration of Melatonin
  Interventions: Drug: Melatonin 20 MG Oral Capsule
- Placebo (Placebo Comparator): The group received standard treatment with the oral administration of Placebo
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Melatonin 20 MG Oral Capsule — The administration of Melatonin 20 mg in addition to neoadjuvant chemotherapy to observe the antioxidant and onco-static effect.
  Arms: Melatonin
Drug: Placebo oral capsule — The administration of placebo capsule in addition to neoadjuvant chemotherapy
  Arms: Placebo

SUMMARY:
Backgrounds

Squamous cell carcinoma of the oral cancer (OSCC) is the sixth most common malignancy. Surgery is the mainstay of treatment for oral cancers. In locally advanced and unresectable oral cancer, surgery presents challenges primarily because the head and neck region have many critical structures that can be damaged by tumor or treatment. Damage to the critical structures can result in significant structural, cosmetic and functional deficits that negatively impact quality of life.

Use of NC was found to achieve resectability in 39% of locally advanced unresectable oral cancers. Patil et al. reported response rate with the three drugs regimen (TPF) for NC was 32% and 27,37% for two drugs regimen (TP). The overall response rate in the TPF group was significantly higher than that in the PF group, both in the induction-chemotherapy phase and after locoregional therapy (33,3% vs 19,9%, p = 0,004). Chemoresistancy has become the challenge in OSCC treatment affecting tumor response to chemotherapy.

Hypoxic microenvironment found in OSCC is marked by the high expression of HIF-1α. CD44 and CD133 as a cancer stem cells marker in head and neck (HNSCC) and miR-210 known as hypoxamiR has been reported to contribute chemoresistancy. As hypoxia inarguably one of the main causes of chemoresistancy, it is agreeable to use melatonin as an antioxidant to reduce the hypoxic condition in tumor microenvironment. Melatonin, a potent endogenous antioxidant agent is proven to have an oncostatic effect, was given in expect to reduce the tumor hypoxic condition so that it would increase the tumor response on NC. Majority of the clinical study use oral melatonin given once daily in 20 mg dose as the minimal dose to yield anti-tumor effects.

The purpose of this study is to prove the effectiveness of melatonin to increase clinical response in locally advanced OSCC patients when treated with NC. The effect of melatonin in reducing tumor hypoxia will be seen through its effect in decreasing the gene expressions of HIF-1α, miR-210, CD44, and CD133.

Methods

Study Design

This study is a double blind, randomized clinical trial using placebo as comparison running from June 2017 to July 2018 . Locally advanced OSSC (stage IVA and IVB) patients that will receive NC were included in the study. Fifty patients treated at two centres (RSCM and RSKD) were randomly allocated into two arms. Twenty-five patients received melatonin combined with three regiment NC (Taxane, Cisplatin, and 5-FU) and the other received placebo with NC. However only 25 out of 50 patients had completed the study protocol (13 patients in melatonin arm and 12 in placebo arm)

Evaluation of Clinical Response

The clinical response were assessed by evaluating pre-treatment and post treatment MRI with the aid of RECIST 1.1. First, it is necessary to estimate the overall tumor burden at baseline (target and non-target lesion) and use this as a comparator for subsequent measurement. The tumor response then being determined according to the definition criteria according to RECIST 1.1, as follows: Complete response (CR) is the disappearance of all target lesions. Partial response (PR) means there is at least 30% decrement in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive disease (PD) means there is at least a 20% increment in the sum of diameters of target lesions or an absolute increment of at least 5 mm. Stable disease (SD) is when there is neither a sufficient shrinkage nor sufficient increment of target lesion. Patients who categorized as PR and CR undergone surgery while those with SD and PD undergone core biopsy.

Genes expression examination

The primer for HIF-1α miR210, CD44, and CD133 genes amplification was design using a Primer Quest Tool IDT software. The total sequence of each gene attained from GenBank data source: National Centre for Biotechnology Information (NCBI). The steps of gene expression examination are RNA isolation, cDNA synthesis, and absolute quantification qPCR. qPCR result was analyzed based on the gene expression concentration compare to the pre-determined standard curve (positive control) of each genes.

Statistical analysis

The data was analysed with statistics software SPSS 20. Saphiro Wilk was used to test data normal distribution. Data with normal distribution and with p > 0,05 presented in mean +- standard deviation (SD). Data with abnormal data distribution presented in median (minimal and maximal value). The statistical difference of gene concentration level (numerical data) between melatonin and placebo was analysed using normality test of Saphiro Wilk. Data with normal distribution was tested using unpaired-T test, while data with abnormal distribution was tested using Mann Whitney. Statistically significant different stated as p < 0,05.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with locally advanced oral squamous cell carcinoma
2. Patients with locally advanced oral squamous cell carcinoma who are planned with neoadjuvant chemotherapy
3. Patients with locally advanced oral squamous cell carcinoma who are planned with neoadjuvant chemotherapy who have not received any definitive treatment modalities, including surgical resection and chemoradiation therapy before the study conducted
4. Patients who are willing to sign the informed consent form to be our subject participants
5. Karnofky >50

Exclusion Criteria:

1. Patients who are already treated with definitive therapy for locally advanced oral squamous cell carcinoma
2. Patients who are not eligible to be treated with chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-04 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diani Kartini, MD, Principal Investigator — Indonesia University
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kartini D, Taher A, Panigoro SS, Setiabudy R, Jusman SW, Haryana SM, Abdullah M, Rustamadji P, Purwanto DJ, Sutandyo N, Suroyo I, Siregar BH, Maruli H, Sungkar S. Effect of melatonin supplementation in combination with neoadjuvant chemotherapy to miR-210 and CD44 expression and clinical response improvement in locally advanced oral squamous cell carcinoma: a randomized controlled trial. J Egypt Natl Canc Inst. 2020 Feb 28;32(1):12. doi: 10.1186/s43046-020-0021-0. PMID 32372215

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Melatonin | Placebo
Started | 25 | 25
Completed | 13 | 12
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Groups:
- Melatonin Group: Participants who received Melatonin (treatment arm) who finished study protocol
- Placebo Group: Participants who received Placebo (control arm) who finished study protocol
- Total: Total of all reporting groups
Arm/Group | Melatonin Group | Placebo Group | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Customized [Count of Participants; unit: Participants]
  Less than or equal to 50 years | 5 | 7 | 12
  Greater than 50 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Indonesia | 13 | 12 | 25
Tumor Location [Count of Participants; unit: Participants]
  Tongue | 10 | 9 | 19
  Buccal | 1 | 1 | 2
  Palate | 0 | 1 | 1
  Mandible | 1 | 1 | 2
  Gingiva (Gum) | 1 | 0 | 1
Stage [Count of Participants; unit: Participants] — Stage of patients is performed referring to 8th edition 2017 American Joint Committee on Cancer (AJCC) Staging based on TNM (Primary tumor, Regional lymph nodes, Distant metastasis). Patients with Stage IVa is in general considered to have a better outcome than those of having Stage IVb.
  Participants
    Stage IV A | 12 | 10 | 22
    Stage IV B | 1 | 2 | 3
Keratinized/non-keratinized [Count of Participants; unit: Participants]
  Keratinized | 12 | 6 | 18
  Non-keratinized | 1 | 6 | 7
Differentiation [Count of Participants; unit: Participants]
  Well Differentiated | 5 | 4 | 9
  Moderately Differentiated | 5 | 3 | 8
  Poorly Differentiated | 3 | 5 | 8
Grade [Count of Participants; unit: Participants]
  High Grade | 6 | 11 | 17
  Low Grade | 7 | 1 | 8
Medication adherence [Count of Participants; unit: Participants]
  Strict adherence | 10 | 9 | 19
  Poor adherence | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response as Measured by RECIST 1.1. Criteria
Description: Clinical Response is measured using RECIST 1.1. criteria. CR (Complete response) is defined as disappearance of all target lesion, and pathological lymph node showing reduction of its shortest axis to less than 10 mm. PR (Partial response) is defined as reduction of total target lesion diameter at least by 30%. PD (Progressive disease) is defined as total target lesion diameter increased in size atleast by 20% or 5 mm OR occurence of one new lesion. SD (Stable disease) is defined as absence of reduction or increasing of target lesion. Patients with PR and CR are considered as positive response. Patients with SD and PD are considered as negative response.
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 13 | 12
Participants
  Positive Response | 5 | 5
  Negative Response | 8 | 7

2. Secondary Outcome: Change in Expression of HIF-1⍺ as Measured by qRT-PCR Absolute Quantification
Description: Expression of HIF-1⍺ is measured at the initial period of the study (baseline) and after 3 neoadjuvant chemotherapy cycles are completed using qRT-PCR Absolute Quantification. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 1 Year
Measure: Median (Full Range); unit: Picogram/microliter
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 13 | 12
Picogram/microliter
  Pre-Treatment | 0.018 [0.0030 to 0.142] | 0.0048 [0.0005 to 0.254]
  Post-Treatment | 0.012 [0.0014 to 0.139] | 0.0087 [0.0004 to 0.060]
  Change (Posttreatment - Pretreatment) | -0.008 [-0.131 to 0.085] | 0.0027 [-0.238 to 0.053]

3. Secondary Outcome: Change in Expression of miR-210 as Measured by qRT-PCR Absolute Quantification
Description: Expression of miR-210 is measured at the initial period of the study (baseline) and after 3 neoadjuvant chemotherapy cycles are completed using qRT-PCR Absolute Quantification. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: Picogram/microliter
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 13 | 12
Picogram/microliter
  Pre-Treatment | 162.8 (54.92) | 175.2 (34.3)
  Post-Treatment | 53.8 (16.65) | 53.5 (14.28)
  Change (Posttreatment - Pretreatment) | -109.09 (51.62) | -103.71 (36.24)

4. Secondary Outcome: Change in Expression of CD44 as Measured by qRT-PCR Absolute Quantification
Description: Expression of CD44 is measured at the initial period of the study (baseline) and after 3 neoadjuvant chemotherapy cycles are completed using qRT-PCR Absolute Quantification. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 1 Year
Measure: Median (Full Range); unit: Picogram/microliter
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 13 | 12
Picogram/microliter
  Pre-Treatment | 0.0349 [0.0048 to 0.1440] | 0.0095 [0.0002 to 0.1170]
  Post-Treatment | 0.0115 [0.0003 to 0.2040] | 0.0187 [0.0012 to 0.2780]
  Change (Posttreatment - Pretreatment) | -0.0114 [-0.0994 to 0.1736] | 0.0082 [-0.1109 to 0.2773]

5. Secondary Outcome: Change in Expression of CD133 as Measured by qRT-PCR Absolute Quantification
Description: Expression of CD133 is measured at the initial period of the study (baseline) and after 3 neoadjuvant chemotherapy cycles are completed using qRT-PCR Absolute Quantification. Change was calculated from two time points as the value at the later time point minus the value at the earlier time point.
Time Frame: 1 Year
Measure: Median (Full Range); unit: Picogram/microliter
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 13 | 12
Picogram/microliter
  Pre-Treatment | 1.13 [0.14 to 4.73] | 1.07 [0.04 to 5.64]
  Post-Treatment | 1.42 [0.11 to 2.85] | 1.88 [0.22 to 20.90]
  Change (Posttreatment - Pretreatment) | 0.43 [-3.50 to 1.37] | 0.55 [-2.33 to 18.20]

ADVERSE EVENTS:
Time Frame: 56 Weeks
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 12/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=13) | Placebo (N=12)
Sleep Pattern Disturbance (Nervous system disorders) | 2 | 2
Fatigue (General disorders) | 2 | 3
Headache (Nervous system disorders) | 3 | 1
Decreased Alertness (Nervous system disorders) | 2 | 0
Sleepiness (Nervous system disorders) | 4 | 3
Emotional Changes (Psychiatric disorders) | 2 | 3
Hallucination (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
There is a significant number of participants that are enrolled at the initial period of study but did not complete the whole study protocol due to various reasons, therefore statistical power of this study becomes lowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04137627/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/27/NCT04137627/SAP_001.pdf